CLINICAL TRIAL: NCT01596764
Title: Effects of Extended Release Methylnaltrexone Bromide (150 mg b.i.d.) in Comparison to Extended Release Naloxone Hydrochloride (20 mg b.i.d.) on Loperamide-induced Delay of the Oro-cecal, Whole-gut and Colon Transit Time in Healthy Subjects.
Brief Title: Effects of Methylnaltrexone in Comparison to Naloxone on Loperamide-induced Delay of the Oro-cecal, Whole-gut and Colon Transit Time.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: LOP-MNTX-2011
Record Dates: First submitted 2012-05-07; First posted 2012-05-11 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Intestinal Obstruction
Keywords: whole-gut transit time; oro-cecal transit time; colon transit time; loperamide-induced obstipation; pharmacokinetics; Methylnaltrexone; Naloxone
MeSH Terms: conditions — Intestinal Obstruction | interventions — Loperamide; Sulfasalazine; Naloxone; methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Placebo Comparator): Administration of LOP Placebo (0 h, 12 h, 24 h, 36 h, 48 h), Colon Transit (0 h, 12 h, 24 h, 36 h, 48 h), Placebo (0 h, 12 h, 24 h, 36 h, 48 h) and SSP (48 h). To assess WGT, OCT and CTT under placebo condition.
  Interventions: Drug: Loperamide placebo; Device: Colon Transit; Drug: Sulfasalazine; Drug: Placebo of MNTX and NLX
- Treatment B (Placebo Comparator): Administration of LOP (0 h, 12 h, 24 h, 36 h, 48 h), Colon Transit (0 h, 12 h, 24 h, 36 h, 48 h), Placebo (0 h, 12 h, 24 h, 36 h, 48 h) and SSP (48 h). To assess WGT, OCT and CTT under loperamide-induced obstipation condition.
  Interventions: Drug: Loperamide; Device: Colon Transit; Drug: Sulfasalazine; Drug: Placebo of MNTX and NLX
- Treatment C (Active Comparator): Administration of LOP (0 h, 12 h, 24 h, 36 h, 48 h), Colon Transit (0 h, 12 h, 24 h, 36 h, 48 h), NLX-ER (0 h, 12 h, 24 h, 36 h, 48 h) and SSP (48 h). To describe the effects of repeated-dose naloxone in preventing loperamide-induced delay of WGT, OCT and CTT and measure pharmacokinetics of naloxone.
  Interventions: Drug: Loperamide; Device: Colon Transit; Drug: Sulfasalazine; Drug: Naloxone
- Treatment D (Active Comparator): Administration of LOP (0 h, 12 h, 24 h, 36 h, 48 h), Colon Transit (0 h, 12 h, 24 h, 36 h, 48 h), MNTX-ER (0 h, 12 h, 24 h, 36 h, 48 h) and SSP (48 h). To describe the effects of repeated-dose methylnaltrexone in preventing loperamide-induced delay of WGT, OCT and CTT and measure pharmacokinetics of methylnaltrexone.
  Interventions: Drug: Loperamide; Device: Colon Transit; Drug: Sulfasalazine; Drug: Methylnaltrexone

INTERVENTIONS:
Drug: Loperamide placebo — 200 ml apple juice
  Other Names: LOP Placebo
  Arms: Treatment A
Drug: Loperamide — 20 ml Loperamid-ratiopharm® Lösung (ratiopharm) in 180 ml apple juice containing 4 mg of loperamide hydrochloride (prepared before administration)
  Other Names: LOP
  Arms: Treatment B; Treatment C; Treatment D
Device: Colon Transit — 5 capsules containing radio-opaque markers of different shapes, respectively
Drug: Sulfasalazine — Azulfidine® Tabletten 500 mg (Pharmacia/Pfizer) containing 500 mg immediate release sulfasalazine
  Other Names: SSP
Drug: Placebo of MNTX and NLX — Placebo capsule (hard gelatine capsule containing multiple sugar spheres)
  Other Names: Placebo
  Arms: Treatment A; Treatment B
Drug: Naloxone — Naloxone hydrochloride 20 mg Extended Release Capsule equivalent to 18 mg naloxone (hard gelatine capsule containing a single NLX-ER tablet and multiple sugar spheres)
  Other Names: NLX-ER
  Arms: Treatment C
Drug: Methylnaltrexone — Methylnaltrexone bromide 150 mg extended release capsule equivalent to 122 mg methylnaltrexone (hard gelatine capsule containing multiple MNTX-ER micro tablets)
  Other Names: MNTX-ER
  Arms: Treatment D

SUMMARY:
The purpose of this study is to describe the effects of repeated-dose methylnaltrexone in preventing loperamide-induced delay of whole-gut, oro-cecal and colon transit time and to measure pharmacokinetics of methylnaltrexone and naloxone-3-glucuronide after oral administration of methylnaltrexone and naloxone.

DETAILED DESCRIPTION:
The increasing prevalence of opioid use and consequently, opioid-induced bowel dysfunction has prompted interest in identifying effective treatment options. Until now, the treatment of opioid-induced constipation (OIC) has been viewed as an extension of constipation in general. Traditional therapies for constipation such as bulking agents, stool softeners, stimulant laxatives, and osmotic agents are commonly utilized, but the effects of such therapies are nonspecific and are often generating diarrhea or cramps and some of these drugs cause severe side effects. Furthermore, these conventional measures are sometimes insufficient in some patients, especially those requiring increasing doses of opioids.

Opioid-induced constipation is predominantly mediated by gastrointestinal μ-opioid receptors. Selective blockade of these peripheral receptors might relieve constipation without compromising centrally mediated effects of opioid analgesia or precipitating withdrawal.

Naloxone is a competitive antagonist of opioid receptors inside and outside the central nervous system used as a solution for injection in the treatment of opioid overdose. When administered orally, it can reduce opioid-induced constipation due to a local action in the gut. It has a high first-pass metabolism, which is an advantage as the laxative effect can be achieved due to the local action in the gut without significant antagonism of the narcotic analgesic effect of opioid. In some patients, however, withdrawal symptoms or reduction of analgesia was seen.

Another way to prevent central actions is the use of opioid antagonists which cannot penetrate the blood-brain barrier such as methylnaltrexone and alvimopan. Their antagonism of μ-opioid receptors in the gastrointestinal tract seems to reverse opioid-induced gut hypomotility.

It is assumed that methylnaltrexone after oral administration influences intestinal motility by local blockade of opioid receptors along the luminal surface of the gut. Because methylnaltrexone seems to have an absorption window in the proximal small intestine as caused by lower activity of P-glycoprotein in that region (similar to other quatenary compounds, eg. trospium chloride), immediate release (uncoated) methylnaltrexone is better absorbed form the small intestine and might therefore be less active than the enteric-coated drug.

However, the pharmacokinetic and pharmacodynamic data on oral methylnaltrexone are very preliminarily so far. The data were obtained in rather small groups with inadequate study design (no randomization, no cross-over, lack of sensitive analytical assays etc.) Furthermore, intestinal transit time has been measured using lactulose as a probe compound that has an own laxative effect.

Therefore, the following clinical study was initiated to proof the concept in a controlled clinical trial in healthy subjects, whether extended release methylnaltrexone antagonizes the loperamide induced delay of oro-cecal and whole-gut transit time in comparison to extended release naloxone.

Loperamide is an opioid agonist and acts on the µ-receptors in the myenteric plexus. It does not affect the central nervous system like other opioids. Loperamide significantly prolongs the mouth-to-cecum transit time as evaluated by the lactulose hydrogen breath test. This effect may be antagonized by the concomitant administration of naloxone.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 45 years
* sex: male and female
* ethnic origin: Caucasian
* minimal body weight: 62 kg
* body mass index:> 19 kg/m² and < 27 kg/m²
* good health as evidenced by the results of the clinical examination, ECG, and the laboratory check-up, which were judged by the clinical investigator not to differ in a clinical relevant way from the normal state
* written informed consent

Exclusion Criteria:

* hepatic and renal diseases and/or pathological findings, which might interfere with pharmacokinetics and pharmacodynamics of the study medication
* gastrointestinal diseases and/or pathological findings, which might interfere with pharmacokinetics and pharmacodynamics of the study medication
* drug or alcohol dependence
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day
* positive results in HIV, HBV and HCV screenings
* volunteers who are on a diet which could affect the pharmacokinetics of the drug
* heavy tea or coffee drinkers (more than 1L per day)
* lactation, pregnancy test positive or not performed or women of child-bearing age without safe contraception
* volunteers suspected or known not to follow instructions of the clinical investigators
* volunteers who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* volunteers liable to orthostatic dysregulation, fainting, or blackouts
* participation in a clinical trial during the last 3 months prior to the start of the study
* less than 14 days after last acute disease
* less than 3 months after last blood donation
* any medication within 4 weeks prior to the intended first administration of the study medication which might influence functions of the gastrointestinal tract (e.g. laxatives, metoclopramide, loperamide, antacids, H2-receptor antagonists, proton pump inhibitors)
* any other medication within two weeks prior to the first administration of the study medication, but at least 10-time the half-life of the respective drug (except oral contraceptives)
* intake of grapefruit containing food or beverages within 14 days prior to administration of the study medication
* known allergic reactions to the active ingredients used or to constituents of the study medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Whole-gut transit time (WGT) | up to 7 days after administration of the study medication
  Whole-gut transit time (WGT) was assessed by counting the radio-opaque markers with different shapes (Colon Transit) at different time pints in the feces.
renal clearance (CLR) | Blood sampling at 48, 49, 50, 50.5, 51, 51.5, 52, 52.5, 53, 53.5, 54, 54.5, 55, 55.5, 56, 57, 58, 60, 62, 64 h and urine sampling 48-60 h after administration of study medication
area under the curve of administration window (AUC0-12h) | 48, 49, 50, 50.5, 51, 51.5, 52, 52.5, 53, 53.5, 54, 54.5, 55, 55.5, 56, 57, 58, 60, 62, 64 h after administration of study medication
maximum concentration at steady state (Css max) | 48, 49, 50, 50.5, 51, 51.5, 52, 52.5, 53, 53.5, 54, 54.5, 55, 55.5, 56, 57, 58, 60, 62, 64 h after administration of study medication
minimum concentration at steady state (Css min) | 48, 49, 50, 50.5, 51, 51.5, 52, 52.5, 53, 53.5, 54, 54.5, 55, 55.5, 56, 57, 58, 60, 62, 64 h after administration of study medication
average concentration of administration interval (Cav) | 48, 49, 50, 50.5, 51, 51.5, 52, 52.5, 53, 53.5, 54, 54.5, 55, 55.5, 56, 57, 58, 60, 62, 64 h after administration of study medication
time of maximum concentration (Tmax) | 48, 49, 50, 50.5, 51, 51.5, 52, 52.5, 53, 53.5, 54, 54.5, 55, 55.5, 56, 57, 58, 60, 62, 64 h after administration of study medication

SECONDARY OUTCOMES:
Oro-cecal transit time (OCT) | 48, 49, 50, 50.5, 51, 51.5, 52, 52.5, 53, 53.5, 54, 54.5, 55, 55.5, 56, 57, 58, 60, 62, 64 h after first administration of study medication
  Oro-cecal transit time (OCT) was defined as the first appearance of sulfapyridine in the plasma (cut of >100 ng/ml) after oral administration of 500 mg sulfasalazine immediate release tablets.
Colon transit time (CTT) | up to 7 days after administration of the study medication
  Colon transit time (CTT) was derived as the difference WGT minus OCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Ernst-Moritz-Arndt-University Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany